CLINICAL TRIAL: NCT07026461
Title: Right-sided 1-Hz Repetitive Transcranial Magnetic Stimulation (rTMS) Versus Left-sided Intermittent Theta Burst Stimulation (iTBS) in Patients With Depression. -a Randomized Non-inferiority Trial
Brief Title: Right-sided 1-Hz Repetitive Transcranial Magnetic Stimulation (rTMS) Versus Left-sided Intermittent Theta Burst Stimulation (iTBS) in Patients With Depression
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.1; CIV-ID 23-06-043272 (Other: Swedish Medical Product Agency)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder; Depression Bipolar
Keywords: rtms; itbs; repetitive transcranial magnetic stimulation; randomized controlled trial; intermittent theta-burst stimulation
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- right-sided rTMS (Experimental): right-sided inhibitory 1 Hz repetitive transcranial magnetic stimulation
  Interventions: Device: repetitive transcranial magnetic stimulation
- left-sided iTBS (Active Comparator): left-sided intermittent theta burst stimulation
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive brain stimulation technique that uses pulsed magnetic fields to activate or suppress specific brain regions. It is used to treat various conditions, including major depressive disorder, by inducing small electrical currents that stimulate nerve cells.
  Other Names: rTMS
  Arms: right-sided rTMS
Device: intermittent theta burst stimulation — Intermittent theta-burst stimulation (iTBS) is a form of transcranial magnetic stimulation (TMS) used to modulate brain activity. It involves delivering brief bursts of magnetic pulses to specific brain regions, typically the left dorsolateral prefrontal cortex (DLPFC)
  Arms: left-sided iTBS

SUMMARY:
Aim: The purpose of the study is to establish the non-inferiority of right-sided inhibitory 1 Hz stimulation compared to left-sided intermittent theta burst stimulation (iTBS) in unipolar and bipolar depression.

Design: A national, non-inferiority, register-based, randomized trial, unmasked, with two treatment arms.

Primary objective: The primary objective is to determine if right-sided inhibitory 1-Hz stimulation to dorsolateral prefrontal cortex (DLPFC) is non inferior to iTBS in treating unipolar and bipolar depression by measuring reduction in Montgomery-Åsberg Depression Rating Scale, self-assessed version (MADRS-S) from baseline to end of treatment.

Secondary objectives: Include testing for differences in:

* Observer rated response according to Clinical Global Impression Scale-Improvement (≥2 point reduction CGI).
* Response to treatment (a decrease of 50% on MADRS-S)
* Self-rated global health measured with the EuroQual-group 5 Dimensions Scale Visual Analogue Scale (EQ-5D-VAS).
* Drop-out from treatment.
* Stimulation site pain measured with the Numerical Rating Scales (NRS).
* Adverse events.
* Admission and suicides within 6 months.
* New treatment course of rTMS or ECT within 6 months
* Remission (score < 11 on the MADRS-S)
* Memory impairment measured with the Comprehensive Psychopathological Rating Scale (CPRS).

Study population: Patients with unipolar or bipolar depression. Sample size: 350 patients.

Inclusion criteria:

* At least 18 years of age at the time of inclusion.
* A clinical diagnosis of unipolar or bipolar depression according to ICD-10.
* Acceptance of rTMS.
* A Swedish personal identity number.
* Capable of giving informed consent.

Exclusion criteria:

• If the investigator judges one of the two treatment protocols inappropriate for the patient.

Inclusion time: 2025-07-01 to 2029-01-01

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of inclusion.
* A clinical diagnosis of unipolar or bipolar depression according to ICD-10.
* Acceptance of rTMS.
* A Swedish personal identity number.
* Capable of giving informed consent.

Exclusion Criteria:

• If the investigator judges one of the two treatment protocols inappropriate for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
reduction in the MADRS-S score | 6 weeks
  reduction in the MADRS-S score from baseline to the end of treatment

SECONDARY OUTCOMES:
Stimulation site pain | 15 minutes
  Stimulation site pain (self-rated by patients using Numerical Rating Scales (NRS)).
CGI-I | 6 weeks
  Professionally determined response according to Clinical Global Impression Scale-Improvement (CGI-I)
Patient rate remission | 6 weeks
  Remission (score < 11 on the MADRS-S)
Patient rated response | 6 weeks
  Response to treatment (a decrease of 50% on MADRS-S)
Self-rated EQ-5D-VAS | 6 weeks
  Self-rated global health measured with the EuroQual-group 5 Dimensions Scale Visual Analogue Scale (EQ-5D-VAS)
Drop-out | 6 weeks
  Drop-out from treatment for any reason within 30 sessions
Adverse events | 6 weeks, follow-up at 6 months
  Adverse events including severe adverse events
Self-rated EQ-5D-VAS at 6-month follow-up | 6 months
  Self-rated global health measured with the EQ-5D-VAS at 6-month follow-up
Self rated remission at 6-month follow-up | 6 months
  Self rated remission (score < 11 on MADRS-S) at 6-month follow-up
Hospital admission | 6 months
  Hospital admissions for depression, hypomanic/manic switch, suicide attempts, and deaths including completed suicides within 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Axel Nordenskjöld, MD, PhD, Study Chair — Region Örebro County, Örebro University; Robert Bodén, MD, PhD, Principal Investigator — Uppsala University, Region Uppsala County
Locations (2):
- Sweden (2):
  - Unit for Brainstimulation, Örebro
  - Unit for Brainstimulation, Uppsala

IPD SHARING:
Plan to Share IPD: No
Data will be available from the corresponding author upon reasonabe request